CLINICAL TRIAL: NCT00852683
Title: The Effects of Peri-Operative Pregabalin on Post-Operative Pain Following Breast Cancer Surgery With Axillary Node Dissection: A Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Peter MacDougall, MD, FRCPC, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDHA-RS/2007-374
Record Dates: First submitted 2008-03-28; First posted 2009-02-27 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer Surgery; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Pregabalin
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — 75 mg twice a day
  Arms: A
Drug: Placebo — 75 mg twice a day
  Arms: B

SUMMARY:
Breast cancer is a devastating disease. Some women with breast cancer undergo surgery to remove the breast and lymph nodes in the axilla (armpit). Unfortunately, surgery of this type is associated with pain both in the days immediately following the operation and in the long term. Pain that continues for more than three months after surgery is known as chronic pain and affects as many as 1/5 to more than ½ of patients having this surgery. Often this pain is of a particular type known as neuropathic pain. There have been studies demonstrating that the intensity of pain after surgery may be related to the likelihood of developing chronic pain. It is important to develop methods to reduce acute pain after breast cancer surgery and to reduce chronic pain for breast cancer survivors.

Pregabalin is a medication used in the treatment of chronic pain. It has been shown to be effective for neuropathic pain. There has also been one study demonstrating its effectiveness in reducing pain after dental extraction. We are interested in determining whether pregabalin taken for 14 days starting the day of surgery will reduce acute (short term) pain and chronic pain from this type of breast cancer surgery.

In order to test ability of pregabalin for the reduction of chronic pain it may be necessary to follow a large number of patients for up to one year after surgery. This may require studying patients in more than one institution. Prior to starting such a large study we are proposing a pilot or preliminary study. This study will follow a smaller group of participants (68) for 6 months. From the pilot study we will determine the effect of pregabalin on acute pain and logistic and statistical information required for the full study. We will randomly assign participants to receive pregabalin or placebo (sugar pills) for twice daily for 14 days starting one hour before surgery. We will monitor the participants' pain at one hour after surgery, 24 hours after surgery, one week, two weeks, three months and six months after surgery. We will also monitor for a number of other parameters such as medication side effects and the need for other pain medications. Recruitment of study participants is expected to take 6-7 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-60 years of age, ASA I-III undergoing breast surgery with axillary dissection for the treatment of breast cancer will be considered eligible for the study.
* Informed consent for the study will be obtained prior to surgery.

Exclusion Criteria:

The following persons will not be considered for inclusion in the study:

* Persons undergoing breast surgery for breast cancer without axillary dissection.
* Persons undergoing cosmetic breast surgery.
* Persons undergoing concurrent breast reconstruction.
* Persons undergoing reconstruction within 12 months of surgery.
* Persons with a history of allergy to gabapentin or pregabalin.
* Persons with a history of allergy to morphine, nonsteroidal antiinflammatory drugs, acetaminophen or oxycodone.
* Persons who are or may be pregnant.
* Persons with a BMI >40.
* Persons with severe organ dysfunction such as liver and renal failure.
* Persons receiving greater than or equal to 30 mg per day of morphine (or equivalent opioid) for pre-existing pain conditions.
* Persons previously on gabapentin or pregabalin within 3 months of surgery.
* Persons with a history of drug abuse. 13) Persons who are unable to communicate in English.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be reduction in Numeric Rating Score (22, 23) at rest (NRS-R) and with movement (NRS-M) 24 hours after surgery. NRS-M is defined as pain with cough or deep inspiration, whichever is greatest. | 24 hours

SECONDARY OUTCOMES:
Incidence of chronic post-mastectomy pain at 3 months defined as persistent pain or discomfort not present prior to surgery and not present as a result of new or recurrent tumour growth. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter MacDougall, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

REFERENCES:
- See also: Capital District Health Authority — http://www.cdha.nshealth.ca